CLINICAL TRIAL: NCT06302816
Title: Comparative Effects of Tupler and Scoop Exercises on Inter-recti-distance, Low Back Pain, Abdominal Strength and Urogynecological Symptoms in Diastasis Recti
Brief Title: Effects of Tupler and Scoop Exercises in Diastasis Recti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0580
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diastasis
Keywords: Diastasis recti abdominis; low back pain; Muscle strength; Pilates-Based Exercises; Static stretching.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUPLER exercises (Experimental)
  Interventions: Other: TUPLER exercises
- SCOOP EXERCISES (Active Comparator)
  Interventions: Other: SCOOP EXERCISES

INTERVENTIONS:
Other: TUPLER exercises — will be conducting tupler exercises, exercises that are designed to target core muscles in order to improve posture, regain core strength and reducing discomfort.
  Each exercise will be repeated 10reps for 3 times on 3 days a week for 8 weeks.
  Arms: TUPLER exercises
Other: SCOOP EXERCISES — will be required to complete scoop exercises basically deals with Pilates which is deep core and hip strengthening and stability through breathing patterns with the utilization of transversus abdominis muscle majorly. In each exercise participant will be asked to hold pelvic floor muscles for 8sec, then relax the muscles and count to 10, repeat I for 10 times each day for 3 days a week for 8weeks. Basic commands about the positing, activation and engagement of core along with breathing control were given to the subjects.
  Arms: SCOOP EXERCISES

SUMMARY:
To compare the effects of tupler and scoop exercises on inter recti distance, low back pain, abdominal strength and urogynecological symptoms in diastasis.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25kg|m^2 to 30kg\m^2or greater
* multiparous women
* Participants included will be 3 months post-partum females
* Caesarean delivery who will have with the presence of DRA >2 finger width and >2cm

Exclusion Criteria:

* patients who had hernia
* trauma to bowel or bladder
* malignancies
* neurologic disease and its associated balance disorders,
* pelvic or abdominal surgery (except for a caesarean section) were considered as the exclusion criteria of this study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — DIASTASIS
Enrollment: 30 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Digital nylon calipers for inter recti distance | 8th week
  Digital nylon calipers for inter recti distance (IRD) used for the evaluatiopn of the DRA using tracing paper can be used preliminary assessment tool as well as a method for documentation of measurements of the inter recti in both males and females above the umbilicus with the abdominal muscles during contraction i.e in hook lying position. Digital Nylon Calipers demonstrated excellent inter-rater (ICC = 0.80 to 0.99) and It is the strongest tool for the assessment of the distasis recti
Numeric pain rating scale | 8th week
  Numeric pain scale is an objective tool for the assessment of pain, rating from 0 to 10 according to the severity of pain. It is categorized as mild(1to3), moderate (4to6) and severe (7to10). It reliability is ICCs for the test-retest reliability were over 0.75
Manual muscle testing for intra-abdominal strength | 8th week
  Manual muscle testing (MMT) is the objective assessment tool for the muscular strength measurement having grading of 0 to 5 according to the muscle response to an active resistance applied passively by some external force that can be therapist's hand. The intra-rater (ICC=0.95) and inter-rater (0.99) reliability (20) . 0 3 4 5 None Fair Good Normal No visible or palpable contraction Full ROM against gravity Full ROM against gravity, moderate resistance Full ROM against gravity, maximal resistance
Short form Pelvic Floor Distress Inventory for Urogynaecological symptoms | 8th week
  Pelvic Floor Distress Inventory (PFDI-20) is a reliable instrument for evaluating the quality of life in women with pelvic dysfunction. They have been translated and validated in many languages. The study was aimed at validating the Estonian translations of the PFDI-20 and PFIQ-7 tools. Intra-class correlation coefficient (ICC) 0.765-0.969, p < 0.001

CONTACTS AND LOCATIONS:
Overall Officials: hina gul gul, Principal Investigator — Riphah International University
Locations (1):
- Innovative Health Concepts, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gluppe S, Engh ME, Bo K. What is the evidence for abdominal and pelvic floor muscle training to treat diastasis recti abdominis postpartum? A systematic review with meta-analysis. Braz J Phys Ther. 2021 Nov-Dec;25(6):664-675. doi: 10.1016/j.bjpt.2021.06.006. Epub 2021 Jul 21. PMID 34391661
- [Background] Tung RC, Towfigh S. Diagnostic techniques for diastasis recti. Hernia. 2021 Aug;25(4):915-919. doi: 10.1007/s10029-021-02469-7. Epub 2021 Jul 27. PMID 34313855
- [Background] Cavalli M, Aiolfi A, Bruni PG, Manfredini L, Lombardo F, Bonfanti MT, Bona D, Campanelli G. Prevalence and risk factors for diastasis recti abdominis: a review and proposal of a new anatomical variation. Hernia. 2021 Aug;25(4):883-890. doi: 10.1007/s10029-021-02468-8. Epub 2021 Aug 6. PMID 34363190
- [Background] Laframboise FC, Schlaff RA, Baruth M. Postpartum Exercise Intervention Targeting Diastasis Recti Abdominis. Int J Exerc Sci. 2021 Apr 1;14(3):400-409. doi: 10.70252/GARZ3559. eCollection 2021. PMID 34055160
- [Background] Kaufmann RL, Reiner CS, Dietz UA, Clavien PA, Vonlanthen R, Kaser SA. Normal width of the linea alba, prevalence, and risk factors for diastasis recti abdominis in adults, a cross-sectional study. Hernia. 2022 Apr;26(2):609-618. doi: 10.1007/s10029-021-02493-7. Epub 2021 Oct 5. PMID 34609664
- [Background] Sułkowski L, Matyja A. Diastasis recti abdominis (DRA): review of risk factors, diagnostic methods, conservative and surgical treatment. 2022.
- [Background] Radhakrishnan M, Ramamurthy K. Efficacy and Challenges in the Treatment of Diastasis Recti Abdominis-A Scoping Review on the Current Trends and Future Perspectives. Diagnostics (Basel). 2022 Aug 24;12(9):2044. doi: 10.3390/diagnostics12092044. PMID 36140446